CLINICAL TRIAL: NCT02221271
Title: Phase III Clinical Trial of NPB-01 in Patients With Guillain-Barré Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nihon Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPB-01-13/C-01
Record Dates: First submitted 2014-08-12; First posted 2014-08-20 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Guillain-Barré Syndrome
MeSH Terms: conditions — Guillain-Barre Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NPB-01 (Experimental)
  Interventions: Drug: NPB-01

INTERVENTIONS:
Drug: NPB-01

SUMMARY:
Patients diagnosed with Guillain-Barré syndrome were confirmed based on the diagnostic criteria for Guillain-Barré syndrome. Patients who meet all inclusion criteria and do not conflict with the exclusion criteria will receive NPB-01 (intravenous immunoglobulin) 400mg/kg/day for five consecutive days.

Patients evaluate the Functional Grade（FG） and Arm Grade（AG） et al.

As a safety endpoint, the safety of NPB-01 will be investigated the occurrence of adverse events by the start of the study treatment.

ELIGIBILITY:
Inclusion Criteria:

1. In principle, patients are able to receive study drug within 2weeks(with limits of 4weeks) from the start of symptoms.
2. Patients with predominant motor neuropathy and Hughes's Functional Grade(FG) is grade4 or grade5(in this regard, if symptoms is progressive, patients with FG is grade3 involve in this study).
3. Patients with plasmapheresis, steroids(in prednisolone equivalent, more than 100mg/day) and immune globulin therapy is no operation for this onset.
4. Patients with greater than or equal to 18 years old at informed consent.

Exclusion Criteria:

1. Patients with history of shock for NPB-01.
2. Patients with history of hypersensitivity for NPB-01.
3. Patients with history of volatile organic solvent abuse, abnormal porphyrin metabolism, history of pharynx or cutaneous diphtheria, plumbism, tephromyelitis, botulism, hysterical paralysis, toxic neuropathy(nitrofurantoin, dapsone, organophosphorous compound), serious diabetic neuropathy,peripheral neuropathy due to HIV,impaired peripheral neuropathy except Guillain-Barré syndrome.
4. Patients with malignancy at informed consent.
5. Patients treated with immune globulin at 8 weeks before informed consent.
6. Patients with IgA deficiency.
7. Patients with impaired liver function.
8. Patients with impaired renal function.
9. Patients with cerebro- or cardiovascular disorders.
10. Patients with high risk of thromboembolism.
11. Patients with hemolytic/hemorrhagic anemia.
12. Patients with decreased cardiac function.
13. Patients with decreased platelet.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
proportion of patients with more than 1grade improvement in the Hughes functional grading scale(FG) relative to baseline at 4weeks. | Baseline,4weeks

SECONDARY OUTCOMES:
days required for 1 grade improvement of the Hughes functional grading scale(FG) | Baseline,1,2,3,4,5,6,7,8,9,10,11,12 weeks
days required for 2 grade improvement of the Hughes functional grading scale(FG) | Baseline,1,2,3,4,5,6,7,8,9,10,11,12 weeks
changes in Hughes functional grading scale(FG) | Baseline,1,2,3,4,5,6,7,8,9,10,11,12 weeks
proportion of patients with more than 1 grade improvement in the Arm Grade(AG) relative to baseline at 4weeks. | Baseline,4weeks
days required for 1 grade improvement of the Arm Grade(AG) | Baseline,1,2,3,4,5,6,7,8,9,10,11,12 weeks
days required for 2 grade improvement of the Arm Grade(AG) | Baseline,1,2,3,4,5,6,7,8,9,10,11,12 weeks
changes in Arm Grade(AG) | Baseline,1,2,3,4,5,6,7,8,9,10,11,12 weeks
changes in manual muscle testing(MMT) | Baseline,1,2,3,4,8,12 weeks
changes in grip strength | Baseline,1,2,3,4,8,12 weeks
changes in activity of daily living(ADL) | Baseline,1,2,3,4,8,12 weeks
changes in electrophysiological findings | Baseline,4,12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Nihon Pharmaceutical Co., Ltd, Osaka, Japan